CLINICAL TRIAL: NCT01803633
Title: Effects of Dairy Fat on Postprandial Inflammation- Phase 2
Brief Title: Determine How Consumption of Dairy Fat as Cheese Influences Inflammation-Phase 2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Dairy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 264297
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Syndrome; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cheese (Experimental): Cheese sandwich plus supplemental beverage will deliver 40% of each participants' energy expenditure and will be made up of 50% of energy as fat, 35% of energy as carbohydrate and 15% of energy as protein. The sandwich will contain medium cheddar cheese and whole wheat bread. The supplemental beverage will contain fruit sorbet, glucose polymer, protein powder, high oleic sunflower oil, high polyunsaturated fatty acids (PUFA) sunflower oil, and canola oil.
  Interventions: Other: Cheddar cheese
- Vegan cheese (Active Comparator): Non-dairy cheese alternative sandwich plus supplemental beverage will deliver 40% of each participants' energy expenditure and will be made up of 50% of energy as fat, 35% of energy as carbohydrate and 15% of energy as protein. The sandwich will contain vegan cheese and whole wheat bread. The supplemental beverage will contain fruit sorbet, glucose polymer, protein powder, cream of tartar, high oleic sunflower oil, high PUFA sunflower oil, and palm oil.
  Interventions: Other: Vegan cheese

INTERVENTIONS:
Other: Cheddar cheese — Tillamook medium cheddar cheese brand
  Arms: Cheese
Other: Vegan cheese — Daiya brand vegan cheese
  Arms: Vegan cheese

SUMMARY:
Phase 2 of this study involves determining how consumption of cheese compared with a non-dairy cheese substitute influences inflammation over a six hour period.

DETAILED DESCRIPTION:
Phase 2 is a randomized crossover study designed to determine how consumption of cheese compared with a non-dairy cheese substitute influences postprandial inflammation in participants who have 2 or more risk factors of metabolic syndrome or BMI ≥ 30.

Eligible participants will arrive to the Western Human Nutrition Research Center (WHNRC) at the University of California (UC) Davis campus on the morning of each test day after a 10-12-hr overnight fast. Upon arrival participants will fill out a questionnaire about their dietary and medication intakes and physical activity for the past 72 hours to ensure compliance. Compliant participants' weight and blood pressure will be measured and a fasting blood draw will be taken before participants consume their test meal (cheese or non-dairy cheese substitute). Participants will only consume this test meal and water freely for the duration of the test day. Blood will be drawn serially at 1, 3 and 6 hours postprandially. Participants will be tested on a second test day two weeks after the first test.

On the second test day, participants' body composition and bone mineral density will be measured by dual x-ray absorptiometry.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Two or more components of metabolic syndrome:

Central obesity (waist circumference greater than 40 inches for men and 35 inches for women); fasting blood triglycerides greater than or equal to 150 mg/dL; plasma HDL cholesterol (Less than 40 mg/dL for men and less than 50 mg/dL for women); blood pressure greater than or equal to 130/85 mmHg; fasting glucose greater than or equal to 100 mg/dL

or

- BMI equal to or greater than 30

Exclusion Criteria:

Metabolic Disorders:

* BMI > 40
* Body weight more than 400 lbs.
* Any immune related diseases such as autoimmune disease, rheumatoid arthritis, asthma,
* Gastrointestinal disorders including Crohn's Disease, colitis, diverticulitis, irritable bowel disease, celiac, malabsorption syndrome
* Cancer
* Known presence of significant metabolic disease which could impact the results of the study (i.e. hepatic, renal disease)
* Type II diabetes
* Use of over-the-counter anti-obesity agents (e.g. containing phenylpropanolamine, ephedrine, and/or caffeine) within the last 12 weeks
* Use of corticoid steroids within the last 12 weeks
* Daily use of anti-inflammatory pain medication
* Self report of eating disorder
* Poor vein assessment determined by WHNRC's phlebotomist

Dietary/supplements:

* Known allergy or intolerance to study food (lactose intolerance, dairy, wheat allergies)
* Vegetarian (defined as abstinence from consumption of eggs, dairy, poultry, beef and pork)
* More than 1 serving of fish per week
* More than 14 grams of fiber per 1000 kcal per day
* Less than 16:1 of total dietary omega 6: Omega 3 ratio
* More than 1% of daily energy as trans fats
* Initiation of anti-inflammatory supplemental fish, krill, flax, borage and primrose seed oils within the last 12 weeks
* Dietary supplements consisting of concentrated soy isoflavones, resveratrol, other polyphenols identified as modulators of inflammation Medications
* Initiation of statin therapy within the last 12 weeks Lifestyle
* More than 10% weight loss or gain during the past 6 months
* Recent initiation (past 4 weeks) of exercise program
* Plan to become pregnant in the next 6 months
* Pregnancy or lactation
* Recent initiation or cessation of hormonal birth control or change in hormonal birth control regimen within the last 12 weeks
* Use of tobacco products
* More than 2 standard alcoholic drinks per day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2013-08-13 (Actual); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Plasma inflammatory mediators | 0, 1, 3, 6 hr postprandial
  Plasma cytokines will be measured using a multi-plex immunoassay and plasma oxylipins will be measured by mass spectroscopy.

SECONDARY OUTCOMES:
Plasma lipid profile | 0, 1, 3, 6 hours postprandial
  Plasma lipids (triglycerides, total cholesterol, LDL-C, HDL-C) will be measured by enzymatic analysis by UC Davis Pathology Lab.
Plasma bone markers | 0, 1, 3, 6 hours postprandial
  Plasma N-terminal telopeptide (NTX), C-terminal telopeptide (CTX) and propeptide of type I collagen (P1NP) will be measured by multi-plex immunoassay.
Urinary metabolites | 0, 1, 3, 6 hours postprandial
  Urinary metabolites will be measured by nuclear magnetic resonance (NMR) spectroscopy.
Plasma glucose | 0, 1, 3, 6 hours postprandial
  Plasma glucose will be measured by enzymatic analysis by UC Davis Pathology Lab.
Plasma lipoprotein size distribution | 0, 1, 3, 6 hours postprandial
  Plasma lipoprotein size distribution and lipoprotein concentrations will be measured by LipoScience using NMR spectroscopy.
Red blood cell functionality | 0, 1, 3, 6 hours postprandial
  Red blood cells isolated from whole blood will be measured for sheer stress using an in-vitro microfluidic assay.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer T. Smilowitz, PhD, Principal Investigator — University of California, Davis; Angela M. Zivkovic, PhD, Principal Investigator — University of California, Davis; Marta Van Loan, PhD, Principal Investigator — ARS USDA WHNRC; J. Bruce German, PhD, Principal Investigator — UC Davis; Bruce D. Hammock, PhD, Principal Investigator — UC Davis
Locations (1):
- USDA Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- [Background] Astrup A, Dyerberg J, Elwood P, Hermansen K, Hu FB, Jakobsen MU, Kok FJ, Krauss RM, Lecerf JM, LeGrand P, Nestel P, Riserus U, Sanders T, Sinclair A, Stender S, Tholstrup T, Willett WC. The role of reducing intakes of saturated fat in the prevention of cardiovascular disease: where does the evidence stand in 2010? Am J Clin Nutr. 2011 Apr;93(4):684-8. doi: 10.3945/ajcn.110.004622. Epub 2011 Jan 26. PMID 21270379
- [Background] Kratz M, Baars T, Guyenet S. The relationship between high-fat dairy consumption and obesity, cardiovascular, and metabolic disease. Eur J Nutr. 2013 Feb;52(1):1-24. doi: 10.1007/s00394-012-0418-1. Epub 2012 Jul 19. PMID 22810464
- [Background] Hostmark AT, Tomten SE. The Oslo health study: cheese intake was negatively associated with the metabolic syndrome. J Am Coll Nutr. 2011 Jun;30(3):182-90. doi: 10.1080/07315724.2011.10719959. PMID 21896876
- [Background] Biong AS, Muller H, Seljeflot I, Veierod MB, Pedersen JI. A comparison of the effects of cheese and butter on serum lipids, haemostatic variables and homocysteine. Br J Nutr. 2004 Nov;92(5):791-7. doi: 10.1079/bjn20041257. PMID 15533268
- [Background] Tholstrup T, Hoy CE, Andersen LN, Christensen RD, Sandstrom B. Does fat in milk, butter and cheese affect blood lipids and cholesterol differently? J Am Coll Nutr. 2004 Apr;23(2):169-76. doi: 10.1080/07315724.2004.10719358. PMID 15047684
- [Result] Demmer E, Van Loan MD, Rivera N, Rogers TS, Gertz ER, German JB, Zivkovic AM, Smilowitz JT. Consumption of a high-fat meal containing cheese compared with a vegan alternative lowers postprandial C-reactive protein in overweight and obese individuals with metabolic abnormalities: a randomised controlled cross-over study. J Nutr Sci. 2016 Feb 9;5:e9. doi: 10.1017/jns.2015.40. eCollection 2016. PMID 27313852
- [Result] Zeng NF, Mancuso JE, Zivkovic AM, Smilowitz JT, Ristenpart WD. Red Blood Cells from Individuals with Abdominal Obesity or Metabolic Abnormalities Exhibit Less Deformability upon Entering a Constriction. PLoS One. 2016 Jun 3;11(6):e0156070. doi: 10.1371/journal.pone.0156070. eCollection 2016. PMID 27258098